CLINICAL TRIAL: NCT04332484
Title: Clinical Validation of the Use of Global Coagulation Tests Like Thromboelastography and Sonoclot in Liver Disease - A Prospective Observational Study.
Brief Title: Global Coagulation Assessment in Cirrhosis and ACLF
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Madhumita Premkumar, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: 586
Record Dates: First submitted 2020-03-30; First posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-04

CONDITIONS: Acute-On-Chronic Liver Failure; Cirrhosis, Liver
Keywords: Sonoclot; Thromboelastography; RoTEM
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute on Chronic Liver Failure: All patients of Acute on chronic liver failure according to CANONIC definition, aged more than 18 years were included. Sonoclot, TEG and conventional coagulation tests were done at baseline and at 72 hours. In case of clinically evident bleeding, Point of care tests were repeated to check for changes.
- Cirrhosis of Liver: All patients with cirrhosis of liver with age more than 18 years were included. Sonoclot, TEG and conventional coagulation tests were done at baseline and at 72 hours. In case of clinically evident bleeding, Point of care tests were repeated to check for changes.

SUMMARY:
Background: Patients with cirrhosis and acute-on-chronic liver failure (ACLF) may have bleeding complications which can lead to increased mortality. Standard coagulation tests (SCTs) like prothrombin time, platelet count and activated partial thromboplastin do not accurately depict in vivo coagulation profile. Point-of-care viscoelastic coagulation testing devices like thrombo-elastography (TEG) and Sonoclot may be better for guiding patient management.

Methods: This prospective observational study compared and validated the point of care (POC) tests and SCTs in 70, 72 and 25 persons with ACLF, decompensated cirrhosis and healthy controls respectively.

ELIGIBILITY:
Inclusion Criteria:

* All patients with Acute on Chronic Liver Failure
* All patients with cirrhosis of Liver

Exclusion Criteria:

* Recent blood or blood component transfusion in last 2 weeks
* HIV infection
* Antiplatelet, anticoagulant or antifibrinolytic therapy
* Patients on Dialysis
* Pregnant females
* Active malignancy in last 5 years
* Chronic heart failure
* Chronic pulmonary disease
* End stage renal disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients of ACLF, Cirrhosis of any etiology and Healthy controls were prospectively enrolled between January 2018 and August 2019.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Validation of TEG and Sonoclot | Day 3
  To clinically validate the comparibility of results obtained from the TEG and Sonoclot instruments

SECONDARY OUTCOMES:
Correlation of Point of care test with standard coagulation tests | Day 3
  To investigate whether variables from TEG or Sonoclot analyses correlated with Standard Coagulation Tests
Correlation of Point of care tests with bleeding event | Day 28
  To assess whether a coagulation defect on TEG or Sonoclot predicts a bleeding event or not.
Correlation of Point of care tests with mortality | 28 days
  To assess whether a coagulation defect on TEG or Sonoclot predicts mortality

CONTACTS AND LOCATIONS:
Locations (1):
- PGIMER, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Premkumar M, Mehtani R, Divyaveer S, Kajal K, Kulkarni AV, Ahmed S, Kaur H, Kaur H, Dhiman R, Duseja A, De A. Clinical Validation of Global Coagulation Tests to Guide Blood Component Transfusions in Cirrhosis and ACLF. J Clin Transl Hepatol. 2021 Apr 28;9(2):210-219. doi: 10.14218/JCTH.2020.00121. Epub 2021 Feb 18. PMID 34007803